CLINICAL TRIAL: NCT02263183
Title: Red Palm Olein and Cardiovascular Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Malaysia Palm Oil Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PD164/12
Record Dates: First submitted 2014-09-22; First posted 2014-10-13 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Cardiovascular Risk Factor
Keywords: Metabolic risk; Abdominally overweight

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- red palm olein(labelled A) (Active Comparator): red palm olein (labelled A)
  Interventions: Dietary Supplement: Red Palm Olein
- palm olein(labelled B)(control) (Placebo Comparator): palm olein(labelled B)(control)
  Interventions: Dietary Supplement: Palm Olein

INTERVENTIONS:
Dietary Supplement: Red Palm Olein — Red Palm Olein contains corresponding fatty acids like Palm Olein except having more phytonutrients (carotenoids and vitamin E)
  Other Names: Carotino
  Arms: red palm olein(labelled A)
Dietary Supplement: Palm Olein — Palm Olein contains corresponding fatty acids like Red Palm Olein except having less phytonutrients (no carotenoids and less vitamin E)
  Other Names: Carotino
  Arms: palm olein(labelled B)(control)

SUMMARY:
Red palm oil is obtained from crude palm oil through a novel low-temperature process. Owing to this special process, RPO possesses a special flavour and aroma, and is rich in phytonutrients that include carotenes, vitamin E, phytosterols, phospholipids, squalene, phenolic acids, flavonoids and co-enzyme Q10. These phytonutrients are the main constituents through which palm oil exhibits its nutritional properties. Among the major health promoting properties are anti-cancer, cardio-protection, anti-angiogenesis, cholesterol inhibition, brain development and neuro-protective properties, antioxidative defence mechanisms, provitamin A activity and anti-diabetes. As red palm oil has variety of phytonutrients and health benefits, the potential of improved cardiovascular health should be considered to understand better and thus treasure more our golden oil.

DETAILED DESCRIPTION:
The oil palm Elaeis guineesis, is the source of palm oil - the 'tropical golden oil'. Malaysia is the world's largest exporter of this golden oil. Triglycerides constitute the major component of crude palm oil, with smaller proportions of diglycerides and monoglycerides. The oil also contains other minor constituents, such as free fatty acids and phytonutrients. This composition determines the oil's physical, chemical and physiological characteristics. In food application, palm oil not only imparts functional properties as a heating medium (as in frying of foods) and in having spreadability (as in formulations for solid fat products like margarines and shortenings), but is also a good source of phytonutrients. Although the phytonutrients constitute only about 1% of its weight in crude palm oil, these are the main constituents through which palm oil exhibits its nutritional properties. Among the major health promoting properties shown to be associated with the various types of phytonutrients present in palm oil are anti-cancer, cardio-protection and anti-angiogenesis, cholesterol inhibition, brain development and neuro-protective properties, antioxidative defence mechanisms, provitamin A activity and anti-diabetes. Red palm oil (RPO) is obtained from crude palm oil through a novel low-temperature process. Owing to this special process, RPO possesses a special flavour and aroma, and is rich in phytonutrients that include carotenes (thus giving the oil a bright red colour), vitamin E, phytosterols, phospholipids, squalene, phenolic acids, flavonoids and co-enzyme Q10.

Little is known about the physiological effects of red palm oil. The link between dietary fats and cardiovascular diseases has always been controversial in the context of palm oil. Narang et al., 2004 demonstrated that the anti-oxidant vitamins in palm olein play a vital role in the protection of the rat's heart against oxidative stress induced by ischemic-reperfusion injury. The unique isomeric position of its fatty acids and the presence of tocotrienols cause the endogenous cholesterol level to drop. Besides palm oil could reduce the risk of arterial thrombosis and atherosclerosis, inhibit endogenous cholesterol biosynthesis, platelet aggregation, and reduce blood pressure. The composition of palm oil with an unsaturated-to-saturated fatty acid ratio close to one and rich in antioxidants vitamins could attenuate the progression of salt-induced hypertension and mortality in rats by modulation of endothelial function and reduction in oxidative stress. In Chinese diet preparation, Zhang et al.,2003 demonstrated that red palm oil is a good source of carotenoids and vitamin E, and it could significantly increase plasma concentration of alpha-carotene, beta-carotene, lycopene and alpha-tocopherol. Following a chronic human study, Scholtz et al., 2004 observed that red palm olein had less detrimental effects on the lipid profile and decreased tissue plasminogen activator antigen as compared to palm olein. As red palm oil has variety of phytonutrients and health benefits, the potential of improved cardiovascular health should be considered to understand better and thus treasure more our golden oil. The present study was designed to investigate the effect of consumption of red palm olein on inflammatory and metabolic risk markers

ELIGIBILITY:
Inclusion Criteria:

* Abdominally obese males and females (waist circumference > 90 cm for male, > 80 cm for female), age between 20-60 years and BMI ≥18.5kgm2 will be recruited.

Exclusion Criteria:

* Medical history of myocardial infarction, angina, thrombosis, stroke, cancer or diabetes
* Blood glucose; >7.0 mmol/L
* Serum triacylglycerol; >4.5 mmol/L
* Serum total cholesterol; >6.5 mmol/L
* Body mass index <18.5 kg/m2
* Current use of antihypertensive or lipid lowering medication
* Alcohol intake exceeding a moderate intake (>28 units per week)
* Breastfeeding or pregnant
* Consume supplement such as herbs and hormone pills
* Smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma Interleukin-6 status | 3 years

OTHER OUTCOMES:
Changes in inflammatory response | 3 years
Changes in endothelial function | 3 years
Changes in lipid profile | 3 years
Changes in plasma antioxidant status | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Radhika Loganathan, Masters, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- Malaysia Palm Oil Board, Kajang, Selangor, Malaysia

REFERENCES:
- [Result] Bayorh MA, Abukhalaf IK, Ganafa AA. Effect of palm oil on blood pressure, endothelial function and oxidative stress. Asia Pac J Clin Nutr. 2005;14(4):325-39. PMID 16326639
- [Result] Choo YM, Ng MH, Ma AN, Chuah CH, Hashim MA. Application of supercritical fluid chromatography in the quantitative analysis of minor components (carotenes, vitamin E, sterols, and squalene) from palm oil. Lipids. 2005 Apr;40(4):429-32. doi: 10.1007/s11745-006-1400-6. PMID 16028723
- [Result] Edem DO. Palm oil: biochemical, physiological, nutritional, hematological, and toxicological aspects: a review. Plant Foods Hum Nutr. 2002 Fall;57(3-4):319-41. doi: 10.1023/a:1021828132707. PMID 12602939
- [Result] Loganathan R Jr, Selvaduray KR, Nesaretnam K, Radhakrishnan AK. Health promoting effects of phytonutrients found in palm oil. Malays J Nutr. 2010 Aug;16(2):309-22. Epub 2010 Aug 15. PMID 22691935
- [Result] Narang D, Sood S, Thomas MK, Dinda AK, Maulik SK. Effect of dietary palm olein oil on oxidative stress associated with ischemic-reperfusion injury in isolated rat heart. BMC Pharmacol. 2004 Nov 9;4:29. doi: 10.1186/1471-2210-4-29. PMID 15535879
- [Result] Scholtz SC, Pieters M, Oosthuizen W, Jerling JC, Bosman MJ, Vorster HH. The effect of red palm olein and refined palm olein on lipids and haemostatic factors in hyperfibrinogenaemic subjects. Thromb Res. 2004;113(1):13-25. doi: 10.1016/j.thromres.2004.02.004. PMID 15081561
- [Result] van Jaarsveld PJ, Benade AJ. Effect of palm olein oil in a moderate-fat diet on low-density lipoprotein composition in non-human primates. Asia Pac J Clin Nutr. 2002;11 Suppl 7:S416-23. doi: 10.1046/j.1440-6047.11.s.7.2.x. PMID 12492628
- [Result] Volek JS, Phinney SD, Forsythe CE, Quann EE, Wood RJ, Puglisi MJ, Kraemer WJ, Bibus DM, Fernandez ML, Feinman RD. Carbohydrate restriction has a more favorable impact on the metabolic syndrome than a low fat diet. Lipids. 2009 Apr;44(4):297-309. doi: 10.1007/s11745-008-3274-2. Epub 2008 Dec 12. PMID 19082851
- [Result] Zhang J, Wang CR, Xue AN, Ge KY. Effects of red palm oil on serum lipids and plasma carotenoids level in Chinese male adults. Biomed Environ Sci. 2003 Dec;16(4):348-54. PMID 15011966